CLINICAL TRIAL: NCT00222105
Title: Doxil® (Pegylated Liposomal Doxorubicin), Dexamethasone Plus Thalidomide (Ddt) in Previously Untreated Multiple Myeloma: A Study Evaluating Efficacy, Toxicity, Harvest Yield and Quality of Life
Brief Title: A Study Evaluating Efficacy, Toxicity, Harvest Yield and Quality of Life
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Doxil
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — liposomal doxorubicin; Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Doxil, Thalidomide, Dexamethasone
  Interventions: Drug: Doxil; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Doxil — Doxil 40 mg/m2 IV day 1
  Other Names: pegylated liposomal doxorubicin
Drug: Thalidomide — 50-100 mg day 1-28
  Other Names: thalidomid
Drug: Dexamethasone — Dexamethasone 40 mg day 1-4 and 15-18
  Other Names: decadron

SUMMARY:
Four monthly treatments with pegylated liposomal doxorubicin, thalidomide and dexamethasone for newly diagnosed myeloma patients as induction therapy prior to high dose chemotherapy and autologous stem cell transplant.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable hematological malignancy of plasma cell origin. Plasma cell clonality and dysfunctional immunoglobulin production characterize the disease. The consequences of abnormal plasma cell growth are manifested by a myriad of symptoms and signs that often have significant impact on the patient's quality of life. These include pancytopenia secondary to predominant distribution of tumor cells within the bone marrow along with many other effects.

This study is focused on the efficacy of Doxil® (pegylated liposomal doxorubicin) with low dose Dexamethasone and Thalidomide (Ddt) in previously untreated patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active, symptomatic multiple myeloma without prior chemotherapy:
* Durie-Salmon Stage II-III A/B
* Stage I patients with at least 2 of the poor prognostic indicators may be eligible.
* Patients with plasma cell leukemia
* Non-secretory multiple myeloma patients are eligible
* Patients between the ages of 18 and 75 years old
* Female Patients of child bearing age (up to age 50) who are not pregnant and agree to use two adequate birth control methods during the study and at least six months after treatment unless patient has undergone hysterectomy or has been in menopause for 2 years.
* Patients with Southwest Oncology Group (SWOG) performance status of 3 or better
* Patients who have received prior lower dose Dexamethasone Therapy (ie. 4 mg QID) as adjunct to radiation therapy for cord compression may be eligible
* All patients must have a MUGA scan indicating a left ventricular ejection fraction (LVEF) of greater than or equal to 50% within 42 days prior to registration
* Must be able to understand English.
* Must be willing and eligible to sign up for the STEPS program

Exclusion Criteria:

* Nursing mothers or women who are pregnant
* Patients with a history of hypersensitivity reaction to doxorubicin or agents in Doxil®
* Patients with previous malignancies at other sites except surgically treated nonmelanomatous skin cancers, prostate cancer or superficial cervical cancers, or other cancer from which the patient had been disease free for 5 or more years.
* History of mediastinal radiation for any reason
* History of receiving prior anthracyclines
* Patients with uncontrolled medical problems such as diabetes mellitus, cardiac, pulmonary, hepatic, and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma
* Myocardial infarction within 6 months of enrollment in the study.
* Major surgery within 4 weeks of enrollment.
* Patients previously treated or receiving other treatment for multiple myeloma other than lower doses dexamethasone as adjunct to radiotherapy
* Pre-existing peripheral neuropathy
* Patients with previously diagnosed malabsorption syndromes or anatomical abnormalities of the gastrointestinal tract that result in malabsorption syndromes.
* Patients with a history of cardiac disease, defined as New York Heart Association Class II or greater, or clinical evidence of congestive heart failure.
* Patients with psychiatric or central nervous systems disorders interfering with compliance of orally administered medication.
* Patients currently receiving anticoagulant therapy for venous thromboembolic episode or other hypercoagulable states.
* Patients who are unable to understand the English language.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-11; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delva Deauna-Limayo, MD, Principal Investigator — University of Kansas Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Doxil, Thalidomide, Dexamethasone
  Doxil: Doxil 40 mg/m2 IV day 1
  Thalidomide: 50-100 mg day 1-28
  Dexamethasone: Dexamethasone 40 mg day 1-4 and 15-18
Period: Overall Study
Arm/Group | Arm 1
Started | 25
Completed | 11
Not Completed | 14
Not completed — Removed due to wrong diagnosis | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 8
Not completed — Treatment delays | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 61 [49 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response rate after completion of first cycle. Measured as the proportion of subjects who have a partial response (PR) or complete response (CR), represented as the overall response rate (ORR). SWOG/IBMTR (Southwest Oncology Group/International Blood and Marrow Transplant Research) criteria utilized to determine multiple myeloma response rates.
Time Frame: At End of Cycle 1, 28 Days
Population: Five subjects did not complete first cycle.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 20
percentage of participants | 95

2. Secondary Outcome: Toxicity
Description: Count of Participants with adverse events.
Time Frame: End of study, up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 25
Participants | 10

ADVERSE EVENTS:
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=25)
Infection (Infections and infestations) | 5 (5)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes